CLINICAL TRIAL: NCT03921216
Title: Cholesterol Metabolism in Plasma and Interstitial Fluid Among Subjects Undergoing Hemodialysis.
Status: Suspended | Type: Observational
Why Stopped: Covid19
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Rudling, Professor, Karolinska University Hospital
Other Study IDs: CKDIC2
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathies; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, interstitial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Diabetic nephropathy, on hemodialysis
- Chronic kidney disease, on hemodialysis: Chronic kidney disease of other causes than Diabetes.
- Chronic kidney disease, predialysis: Renal outpatients at Nephrology Unit, Karolinska University Hospital Huddinge
- Diabetic nephropathy, predialysis: Renal outpatients at Nephrology Unit, Karolinska University Hospital Huddinge

SUMMARY:
Because the atherosclerosis process partly occur in the intercellular space of the vessel wall, the determination of the constitution of lipoproteins in the interstitial fluid may expand the knowledge about the atherosclerosis process and lead to a better understanding of what constitutes the increased risk of developing cardiovascular disease in patients with chronic diseases. The investigators hypothesize that the apoB-containing particles in T2D patients are more susceptible to be retained or consumed in the intercellular compartment, which in turn could be one explanation for the elevated risk of atherosclerosis. The investigators hypothesise that with the progression of chronic kidney disease this process is further increased. Patients undergoing dialysis are known to have a very high risk of cardiovascular disease. The investigators now want to study the cholesterol metabolism in interstitial fluid in subjects undergoing hemodialysis because of diabetic nephropathy and in subjects undergoing hemodialysis because of chronic kidney disease of other causes.

ELIGIBILITY:
Inclusion Criteria:

Diabetic nephropathy, because of type 2 diabetes, undergoing hemodialysis and subjects with chronic kidney disease of other causes undergoing hemodialysis.

Exclusion Criteria:

* Active infection that increases the risk of secondary infection in the skin where the vesicles containing interstitial fluid have been emptied of interstitial fluid with a fine needle and the bladder roof is intact.
* Treatment with Warfarin due to increased risk of Calciphylaxis (calcific uremic arteriolopathy, CUA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic nephropathy, because of type 2 diabetes, undergoing hemodialysis and subjects with chronic kidney disease of other causes undergoing hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Interstitial fluid-to-serum ratio for LDL cholesterol | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mats Rudling, Principal Investigator — Karolinska Institutet
Locations (1):
- Dialysis Unit, M87-89, Karolinska University Hospital, Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No